CLINICAL TRIAL: NCT06851013
Title: Multisite Precision Study for the SpinChip High-sensitivity Cardiac Troponin I (SpinChip Hs-cTnI) Test
Brief Title: SpinChip Hs-cTnI Multisite Precision
Acronym: HEAT-1
Status: Completed | Type: Observational
Sponsor: SpinChip Diagnostics ASA (Industry)
Collaborators: Aurevia (Industry)
Responsible Party: Sponsor
Other Study IDs: Design Protocol-03821; CIV-NO-24-09-049195 (Other: EUDAMED)
Record Dates: First submitted 2025-02-19; First posted 2025-02-28 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: Acute Myocardial Infarction; High-sensitive; Point of care; Troponin I; Near-patient test; Heart attack; Diagnostic accuracy
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Li-heparin plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: SpinChip hs-cTnI — SpinChip Platform, consisting of the SpinChip hs-cTnI test (self-contained cartridge) and SpinChip Analyzer (instrument)

SUMMARY:
During a heart attack, the protein troponin I is released from the heart muscle into the bloodstream. Measurements of cardiac troponin in blood are used as an aid in the diagnosis of heart attack. The SpinChip hs-cTnI test is a new high-sensitive test for measuring the amount of cardiac troponin I in the bloodstream as an aid in the diagnosis of heart attack.

The purpose of this study is to establish the precision of the SpinChip hs-cTnI test when using Li-Heparin plasma and whole blood samples in the hands of the intended user in the intended use setting at multiple sites.

DETAILED DESCRIPTION:
Cardiac troponins are widely used as a biomarker to aid in the diagnosis of acute myocardial infarction (AMI). These structural proteins are essential in regulating contraction in cardiac muscle cells, and they are sensitive and specific biochemical markers of myocardial damage.

During a heart attack, cardiac muscle cells are injured and release the cardiac marker troponin I (cTnI) into the bloodstream. High-sensitive troponin tests may detect the increase of cardiac troponin in blood within hours after the symptoms of a heart attack has started.

The SpinChip high-sensitivity cardiac troponin I (hs-cTnI) test is a new high-sensitive test for measuring troponin I in blood samples, and the analysis may be performed close to the patient (near-patient test). The results may be obtained within 10 minutes, compared to approximately 1 hour for normal laboratory analysis.

The SpinChip Platform consists of the SpinChip hs-cTnI test and the SpinChip Analyzer and may be used at the emergency department to evaluate patients presenting with symptoms of acute myocardial infarction (chest pain). The test can use blood from finger prick or venous blood samples, either as whole blood or separated into plasma.

This multisite prospective, observational, non-randomized validation study will establish the repeatability, within-laboratory precision and reproducibility of the SpinChip hs-cTnI test for Li-Heparin plasma and repeatability for Li-Heparin whole blood samples. Potential subjects will be identified based on clinical cardiac troponin levels obtained from medical records at the individual study site.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide signed written informed consent
* Subjects >18 years old
* Clinical cTn concentrations available

Exclusion Criteria:

* Cognitive impairment precluding informed consent
* Self-reported pregnancy
* General clinical condition that affects the patient in a major way and the patient is considered to be in an unstable clinical condition
* Previously included in the study with a sample within the required concentration ranges for the SpinChip hs-cTnI test
* No venous blood sample collected for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized, adult subjects with known cTn values obtained from medical records. The study population will be recruited from two clinical sites in Norway.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Precision of the SpinChip hs-cTnI test using Li-heparin plasma and whole blood samples | 1 day
  Calculation of repeatability, within-laboratory precision and reproducibility of the SpinChip hs-cTnI test using cTnI results obtained from analysis of Li-Heparin plasma. Calculation of repeatability of the SpinChip hs-cTnI test using cTnI results obtained from analysis of Li-Heparin whole blood.

SECONDARY OUTCOMES:
Precision of the recommended commercially available control material | 1 day
  Calculation of repeatability, within-laboratory precision and reproducibility of the SpinChip hs-cTnI test using cTnI results obtained from analysis of commercial control material
Incidence of AEs, ADEs and DDs | 1 day
  Evaluate safety of the SpinChip Platform, as measured by adverse events (AEs), adverse device effects (ADEs) and device deficiencies (DDs).

CONTACTS AND LOCATIONS:
Overall Officials: Hlge Røsjø, MD/Professor, Principal Investigator — Akershus University Hospital, Akershus Clinical Research Center (ACR), Norway
Locations (3):
- Norway (3):
  - Akershus University Hospital, Akershus Clinical Research Center (ACR), Lørenskog, Akershus
  - Vestre Viken Bærum Hospital, Sandvika, Akershus
  - SpinChip Diagnostics, Oslo, Oslo County

IPD SHARING:
Plan to Share IPD: No